CLINICAL TRIAL: NCT02363309
Title: Palmitate Breath Test to Assess Fatty Acid Oxidation in Non Alcoholic Fatty Liver Disease
Brief Title: Palmitate Breath Test to Assess Fatty Acid Oxidation in Non Alcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150080; 15-DK-0080
Record Dates: First submitted 2015-02-13; First posted 2015-02-16 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Fatty Liver
Keywords: 13C; Fatty Liver; Acetate; Breath Tests; Palmitate
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteers: Subjects without liver disease or metabolic syndrome
- NAFLD subjects: Subjects with Non-Alcoholic Fatty Liver Disease
- non-NAFLD metabolic syndrome: Subjects who have metabolic syndrome but do not have Non-Alcoholic Fatty Liver Disease

SUMMARY:
Background:

- Non-alcoholic fatty liver disease (NAFLD) is a common cause of abnormal liver tests. It is closely linked to health problems like obesity and diabetes. Researchers want to use a breath test to measure the metabolism of fatty acids and learn more about the causes of disease. They will compare the results between people who do and do not have NAFLD. They will also repeat the test in people with NAFLD after treatment to see improvement.

Objectives:

- To measure the metabolism of fatty acids and compare them between people who do and do not have NAFLD, and people with NAFLD before and after treatment.

Eligibility:

* People age 21 and older with NAFLD
* Healthy volunteers
* non-NAFLD metabolic syndrome

Design:

* Participants will be screened with medical history, physical exam, and fasting blood tests.
* Participants will fast overnight.
* Participants will sit in a comfortable chair. They will relax for 15 minutes. Then a narrow plastic tube will be put under their nostrils. It will be connected to a breath test device.
* Participants will drink palmitate or acetate in a heated liquid meal (Ensure). Palmitate is a fatty acid and acetate is a small molecule that is a building block for fatty acids. Both palmitate and acetate are natural compounds that are in our body and our food.
* Participants will sit for 6 hours. They can read, watch television, work on a computer, or other relaxed activity. The air they breathe out from their nose will be collected and analyzed. They may take a bathroom break after 3 hours. They may drink water after 3 hours.
* Participants will get a meal after the test.
* Participants will have another visit at least 1 week later. They will repeat the test with the other compound (acetate of palmitate).
* Participants may be asked to repeat a test to study the result of a change like weight loss or medicine. Thus, participation can last from 1 week to several years.

DETAILED DESCRIPTION:
NAFLD is the most common cause for liver enzyme abnormalities in the western world. It is estimated to affect approximately 30% of the US population and is closely associated with the metabolic syndrome and insulin resistance. Dysregulation of fatty acid metabolism and abnormal function of the adipose tissue is thought to be a major feature of insulin resistance and NAFLD. Whether fatty acid oxidation is also dysregulated in patients with NAFLD is unclear. In this study we aim to measure total-body fatty acid oxidation of an oral fat load using the BreathID breath test device and a meal containing 13C-labeled palmitate. Results will be compared between patients with NAFLD, healthy controls and patients with metabolic syndrome but not NAFLD, as well as within NAFLD patients before and after therapeutic interventions.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. General Inclusion Criteria for all subjects:

1. Age above 21 years, male or female.
2. Estimated average alcohol consumption < 30 g/d for men or < 20 g/d for women in the 6 months prior to enrollment and no binge-drinking behavior.

B. Inclusion Criteria for NAFLD:

1. Clinical suspicion of NAFLD, defined by a liver biopsy result consistent with NAFLD or the presence of at least two of the following criteria:

   1. Suggestion of liver fat by an imaging study (ultrasound, CT scan, MRI or MR spectroscopy) performed in the 6 months prior to enrollment.
   2. Elevated aminotransferase levels (ALT > 31 U/L for men or > 19 U/L for women, or AST > 30 U/L) on at least two occasions in the 6 months preceding enrollment.
   3. Presence of the metabolic syndrome, defined according to the modified AHA/NCEP criteria30 as the presence of at least three of:

      * Abdominal obesity, defined as waist circumference > 102 cm for men or > 88 cm for women
      * Elevated triglycerides (> 150 mg/dL) or the use of medication to lower triglycerides
      * Reduced HDL cholesterol (< 40 mg/DL for men or < 50 mg/dL for women)
      * Elevated blood pressure (> 135/80 mmHg) or use of medication for hypertension
      * Elevated fasting glucose levels (> 100 mg/dL) or use of antidiabetic medication

   For the purpose of inclusion, the presence of overt diabetes mellitus type 2 will be considered equivalent to the presence of the metabolic syndrome, even if the other criteria are absent.

   For the longitudinal analysis, inclusion criteria:
2. Enrolled in 13-DK-0002

   or
3. Non-alcoholic liver disease subjects treated off-protocol with lifestyle intervention or vitamin E treatment.

C. Inclusion Criteria for non-NAFLD metabolic syndrome:

1. Evidence of metabolic syndrome as defined in NAFLD criterion 1.c.
2. Normal transaminases (ALT less than or equal to 31 U/L for men or less than or equal to19 U/L for women, or AST less than or equal to 30 U/L) at screening
3. Absence of liver fat by imaging or liver biopsy within 6 months of screening with no (or trace) liver fat

D. Inclusion criteria for healthy volunteers

1. No history of known liver disease
2. Not on any regular systemic medications (with the exception of oral contraceptives)
3. BMI less than or equal to 25 kg/m2
4. Non diabetic
5. Normal ALT and fasting glucose

EXCLUSION CRITERIA:

1. Disorders leading to CO2 retention or significant respiratory abnormalities such as severe congestive heart failure, severe pulmonary hypertension or severe chronic obstructive lung disease.
2. Disorders interfering with substrate absorption such as gastric bypass surgery, malabsorption disorders, use of orlistat or bile acid sequestrants, or extensive small bowel resection.
3. Pregnancy or lactation
4. Inability to remain seated for the duration of the test.
5. Inability to understand and give informed consent
6. Chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV). Patients who were treated successfully for HCV and achieved sustained virological response can be eligible for enrollment > 18 months after treatment cessation. Patients who are inactive carriers of HBV (HBV DNA < 1000 copies/mL, HBeAg negative, Anti HDV negative) for at least 12 months prior to enrollment are also eligible. Patients receiving antiviral therapy are ineligible.
7. Concomitant liver disease such as autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson s disease, alpha-1 antitrypsin deficiency.
8. Presence of definite or probable drug-induced liver injury. In the case of lipid-lowering, anti-hypertensive or anti-diabetic medications that are suspected to cause elevation of aminotransferases, patients will be eligible if treatment is associated with stable enzyme levels for at least 6 months and inclusion criteria 2a. and 2c. are both present.
9. Treatment with medications known to cause fatty liver disease such as atypical neuroleptics, tetracycline, methotrexate or tamoxifen
10. Diabetic patients requiring insulin treatment
11. Milk or soy protein allergy
12. Uncontrolled hypo/hyperthyroidism

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary clinical and community sample
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2015-03-27 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
Measure rates of fatty acid oxidation in patients with non alcoholic fatty liver disease | End of study
  Differences in rates of fatty acid oxidation in patients with non alcoholic fatty liver disease.

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Rotman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-DK-0080.html